CLINICAL TRIAL: NCT03641378
Title: Multi-Site Randomized Trial of Inpatient Palliative Care for Patients With Hematologic Malignancies Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Inpatient Palliative Care for Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-261; R01CA222014 (NIH)
Record Dates: First submitted 2018-08-14; First posted 2018-08-22 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Stem Cell Transplant
Keywords: Cancer Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient Palliative Care Intervention (Experimental): * Patients and Caregivers will complete baseline self-report assessments at the time of obtaining informed consent
  * Palliative Care Intervention
  * Therapeutic Relationship
    --Develop a strong therapeutic relationship with patients and caregivers
  * Assessment and Treatment of Patient Symptoms
    --Clarify the symptoms the patient will likely experience and offer reassurance about the methods for reporting and treating symptoms
  * Managing Patients and Caregivers Expectations
    --Address early on patients and caregivers' concerns about the trajectory of illness during HCT and treatment side effects
  * Coping with Illness and HCT --Introduce strategies to help improve adjustment (e.g., behavioral, cognitive, and spiritual approaches; accepting illness while maintaining hope; social support)
  Interventions: Other: Palliative Care Intervention
- Transplant Care Alone (Experimental): * Patients and Caregivers will complete baseline self-report assessments at the time of obtaining informed consent.
  * Standard Transplant Care
  Interventions: Other: Standard Transplant Care

INTERVENTIONS:
Other: Palliative Care Intervention — team of clinicians that specialize in the lessening (palliation) of many distressing symptoms
  Arms: Inpatient Palliative Care Intervention
Other: Standard Transplant Care — Standard care per hospital guidelines
  Arms: Transplant Care Alone

SUMMARY:
This research study is evaluating the impact of early involvement of a palliative care team working with the transplant oncology team will have on the quality of life, symptoms, and mood of patients undergoing stem cell transplantation.

DETAILED DESCRIPTION:
The Participant has a type of blood cancer and will be undergoing stem cell transplantation. Frequently people undergoing stem cell transplantation experience physical and emotional symptoms during the course of their hospitalization for stem cell transplantation. These can be very distressing to both patient and the family members. The study doctors want to know if the early introduction of a team of clinicians that specialize in the lessening (palliation) of many of these distressing symptoms may improve the participant overall care.

This team of clinicians is called the palliative care team and they focus on ways to improve the participant pain and other symptom management (nausea, fatigue, shortness of breath, anxiety, etc.) and to assist the participant and the participant's family in coping with the emotional and social issues associated with your diagnosis. The team consists of physicians and advance practice nurses who have been specially trained in the care of patients facing serious illness.

The main purpose of this study is to compare two types of care - standard transplant oncology care and standard transplant oncology care with early involvement of palliative care clinicians to see which is better for improving the experience of patients and families with blood cancers undergoing stem cell transplantation.

The purpose of this research study is to find out whether introducing patients and families undergoing stem cell transplantation to the palliative care team that specializes in symptom management can improve the physical and psychological symptoms that patients and families experience during hospitalization for stem cell transplantation.

The study will use a series of questionnaires to measure the participant and the participant 's caregivers' quality of life, physical symptoms, and mood. Study questionnaires will be completed in the hospital or clinic with assistance provided as need.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria

* adult patients (≥ 18 years) with hematologic malignancy admitted for autologous or allogeneic HCT.
* ability to read and respond to questions in English or Spanish or to complete questionnaires with assistance from an interpreter.

Caregiver Eligibility Criteria:

* adult (≥ 18 years) relative or a friend of a patient who agrees to participate in the study whom the patient identified as living with them or having in-person contact with him or her at least twice per week.
* ability to read and respond to questions in English or Spanish or to complete questionnaires with the assistance of an interpreter.

Exclusion Criteria:

Patient Exclusion Criteria

* Patients undergoing HCT for benign hematologic conditions
* Patients undergoing outpatient HCT.
* Patients with psychiatric or cognitive conditions which the treating clinicians believes prohibits compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Jawahri A, LeBlanc TW, Kavanaugh A, Webb J, Fausto J, Traeger L, Greer JA, Jackson V, Horick N, Rabideau DJ, Fenech A, Newcomb R, Ufere NN, Caruso E, Pepper J, DeFilipp Z, Chen YB, Lee SJ, Temel JS. Multisite Randomized Trial of Inpatient Palliative Care Intervention for Patients Undergoing Hematopoietic Stem Cell Transplantation. J Clin Oncol. 2025 Aug 20;43(24):2700-2711. doi: 10.1200/JCO-25-00378. Epub 2025 Jun 23. PMID 40549982
- [Derived] Newcomb R, Amonoo HL, Kavanaugh AR, Wharton KC, Rowland M, Fausto J, Webb J, Jackson V, Greer JA, Temel JS, Lark P, Rabideau DJ, O'Brien K, LeBlanc TW, Lee SJ, El-Jawahri A. Factors associated with early quality-of-life response to palliative care during hematopoietic cell transplantation. Blood Adv. 2025 May 13;9(9):2033-2043. doi: 10.1182/bloodadvances.2024014574. PMID 39908568
- [Derived] Yang D, Newcomb R, Kavanaugh AR, Khalil D, Greer JA, Chen YB, DeFilipp Z, Temel J, Lee SJ, LeBlanc TW, El-Jawahri A. Protocol for multi-site randomized trial of inpatient palliative care for patients with hematologic malignancies undergoing hematopoietic stem cell transplantation. Contemp Clin Trials. 2024 Mar;138:107460. doi: 10.1016/j.cct.2024.107460. Epub 2024 Jan 26. PMID 38280483
- [Derived] Newcomb R, Amonoo HL, Nelson AM, Choe J, Holmbeck K, Nabily A, Lee SJ, LeBlanc TW, El-Jawahri A. Coping in patients with hematologic malignancies undergoing hematopoietic cell transplantation. Blood Adv. 2024 Mar 26;8(6):1369-1378. doi: 10.1182/bloodadvances.2023011081. PMID 38181820

RESULTS

PARTICIPANT FLOW:
Groups:
- Inpatient Palliative Care Intervention Patients: * Patients will complete baseline self-report assessments at the time of obtaining informed consent
  * Palliative Care Intervention entails having patients seen by a palliative care clinician during their hospitalization for HCT at least twice weekly throughout the transplant hospitalization
- Transplant Care Alone Patients: * Patients will complete baseline self-report assessments at the time of obtaining informed consent.
  * Standard Transplant Care
  Standard Transplant Care: Standard care per hospital guidelines
- Inpatient Palliative Care Caregivers: Patients enrolled in the study and randomized to inpatient palliative care can identify a caregiver who is willing to participate in the study. Patients without an eligible caregiver are still eligible to participate.
  Caregivers will receive the palliative care intervention based on the patient assignment. Caregivers will be allowed to attend palliative care visits with the patients.
- Transplant Care Alone Caregivers: Caregivers of patients randomized to transplant care alone will receive standard transplant care offered by the hospital.
Period: Overall Study
Arm/Group | Inpatient Palliative Care Intervention Patients | Transplant Care Alone Patients | Inpatient Palliative Care Caregivers | Transplant Care Alone Caregivers
Started | 180 | 180 | 101 | 85
Completed | 173 | 160 | 87 | 79
Not Completed | 7 | 20 | 14 | 6

BASELINE CHARACTERISTICS:
Groups:
- Inpatient Palliative Care Intervention - Patients: * Patients will complete baseline self-report assessments at the time of obtaining informed consent
  * Patients randomized to the intervention will receive the palliative care intervention during their hospitalization for transplant in addition to standard transplant care. the palliative care intervention entails having palliative care clinicians see patients at least twice weekly during hospitalization for transplant.
- Transplant Care Alone - Patients: * Patients will complete baseline self-report assessments at the time of obtaining informed consent.
  * Standard Transplant Care
  Standard Transplant Care: Standard care per hospital guidelines
- Inpatient Palliative Care - Caregivers: - Caregivers will be randomized based on the patient's randomization. they complete baseline assessment. if the patient is randomized to the palliative care intervention, the caregiver is also considered in this arm. they are permitted to attend the palliative care visits with the patients during hospitalization for transplant.
- Transplant Care Alone- Caregivers: Caregivers complete baseline assessments and are randomized based on the random assignment of the patient. if the patient is randomized to standard transplant care, then the caregiver is randomized to standard transplant care.
- Total: Total of all reporting groups
Arm/Group | Inpatient Palliative Care Intervention - Patients | Transplant Care Alone - Patients | Inpatient Palliative Care - Caregivers | Transplant Care Alone- Caregivers | Total
Number analyzed (Participants) | 180 | 180 | 101 | 85 | 546
Age, Continuous [Mean (Full Range); unit: years] | 55.3 [21 to 76] | 55.5 [19 to 78] | 54.7 [20.8 to 76.8] | 55.1 [18.8 to 77.7] | 55.4 [18.8 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 65 | 78 | 67 | 282
  Male | 108 | 115 | 23 | 18 | 264
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 2 | 0 | 7
  Asian | 8 | 12 | 10 | 3 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 26 | 15 | 7 | 3 | 51
  White | 134 | 142 | 75 | 74 | 425
  More than one race | 6 | 4 | 5 | 3 | 18
  Unknown or Not Reported | 4 | 3 | 2 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Quality of Life (QOL): Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT)
Description: Compare patient QOL using the Functional Assessment of Cancer Therapy- Bone Marrow Transplant (FACT-BMT) scores at week 2 between the study groups Score range 0-164 with higher score indicating better quality of life
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Inpatient Palliative Care Intervention: * Patients and Caregivers will complete baseline self-report assessments at the time of obtaining informed consent
  * Palliative Care Intervention
  * Therapeutic Relationship
    --Develop a strong therapeutic relationship with patients and caregivers
  * Assessment and Treatment of Patient Symptoms
    --Clarify the symptoms the patient will likely experience and offer reassurance about the methods for reporting and treating symptoms
  * Managing Patients and Caregivers Expectations
    --Address early on patients and caregivers' concerns about the trajectory of illness during HCT and treatment side effects
  * Coping with Illness and HCT --Introduce strategies to help improve adjustment (e.g., behavioral, cognitive, and spiritual approaches; accepting illness while maintaining hope; social support)
  Palliative Care Intervention: team of clinicians that specialize in the lessening (palliation) of many distressing symptoms
- Transplant Care Alone: * Patients and Caregivers will complete baseline self-report assessments at the time of obtaining informed consent.
  * Standard Transplant Care
  Standard Transplant Care: Standard care per hospital guidelines
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 173 | 160
score on a scale | 94.69 (22.5) | 90.09 (18.76)

2. Secondary Outcome: Patients' Quality of Life (QOL) Longitudinally: FACT-BMT
Description: Compare patients' QOL using Functional Assessment of Cancer Therapy- Bone Marrow Transplant (FACT-BMT) longitudinally between the study groups Score range 0-164, with higher score indicating better quality of life
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 180 | 180
score on a scale | 107.8 (23.85) | 108.8 (19.64)

3. Secondary Outcome: Patients' Symptom Burden
Description: Compare patients' symptoms using the revised Edmonton Symptom Assessment Scale (ESAS) scores between the study groups score range 0-100 with higher score indicating worse symptom burden
Time Frame: up to 6 months
Population: at week-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 173 | 160
score on a scale | 35.63 (21.51) | 39.86 (20.83)

4. Secondary Outcome: Patients' Fatigue
Description: Compare patients' fatigue using Functional Assessment of Cancer Therapy- Fatigue (FACT-fatigue) scores between the study groups score range from 0-52 with higher scores indicating lower fatigue symptoms
Time Frame: up to 6 months
Population: week-2 analyses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 171 | 158
score on a scale | 28.3 (12.65) | 25.96 (11.91)

5. Secondary Outcome: Patients' Psychological Distress
Description: Compare patients' depression and anxiety symptoms using the Hospital Anxiety and Depression Scale (HADS) between the study groups The HADS consists of two subscales assessing depression and anxiety symptoms, with scores ranging from 0 (no distress) to 21 (maximum distress)
Time Frame: up to 6 months
Population: depression at week-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 170 | 160
score on a scale | 6.17 (7.89) | 6.63 (4.20)

6. Secondary Outcome: Patients' Depression
Description: Compare patients' depression using Patient-Health Questionnaire - 9 (PHQ-9) between the study groups the PHQ-9 score ranges from 0-27, with higher score indicative more depressive symptoms
Time Frame: up to 6 months
Population: depression (PHQ-9) by week-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 169 | 156
score on a scale | 6.70 (5.20) | 7.07 (4.91)

7. Secondary Outcome: Patients' Post-traumatic Stress Symptoms (PTSD)
Description: Compare patients' post-traumatic stress symptoms using the PTSD Checklist- Civilian version (PCL-C) between the study groups PCL-C score ranges from 17-85 with higher scores indicating worse PTSD symptoms
Time Frame: up to 6 months
Population: analyses at week-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 168 | 156
score on a scale | 26.04 (9.37) | 28.17 (10.91)

8. Secondary Outcome: Caregiver QOL: CARGOQOL
Description: Compare caregivers' QOL using caregiver oncology QOL questionnaire (CARGOQOL) scores between the study groups the caregiver oncology QOL questionnaire ranges from 0-116 with higher scores indicating better caregiver QOL.
Time Frame: up to 6 months
Population: at week-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 87 | 79
score on a scale | 73.86 (12.88) | 73.51 (12.53)

9. Secondary Outcome: Caregiver Psychological Distress
Description: Compare caregivers' psychological distress using hospital anxiety and depression scale (HADS) between the study groups the HADS consists of two subscales assessing depression and anxiety symptoms, with scores ranging from 0 (no distress) to 21 (maximum distress)
Time Frame: up to 6 months
Population: caregiver anxiety at week-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 87 | 79
score on a scale | 6.82 (4.24) | 7.84 (9.13)

10. Secondary Outcome: Caregiver Depression
Description: Compare caregivers' depression symptoms using the Patient Health Questionnaire - 9 (PHQ-9) between the study groups the PHQ-9 score ranges from 0-27 with higher scores indicating worse depression symptoms.
Time Frame: up to 6 months
Population: week-2 caregiver depression (PHQ-9)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Palliative Care Intervention | Transplant Care Alone
Number analyzed (Participants) | 87 | 79
score on a scale | 4.64 (4.54) | 4.73 (4.00)

11. Other Pre Specified Outcome: Patient Coping
Description: Compare patient coping using the Brief Cope questionnaire between the study groups We will administer 14 items of the Brief COPE comprising seven subscales (active coping, use of emotional support, positive reframing, acceptance, behavioral disengagement, denial, and self-blame). Higher scores on each subscale indicate more use of that particular coping strategy.
Time Frame: up to 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Caregiver Coping
Description: compare caregiver coping (Brief Cope) between the study groups. We will administer 14 items of the Brief COPE comprising seven subscales (active coping, use of emotional support, positive reframing, acceptance, behavioral disengagement, denial, and self-blame). Higher scores on each subscale indicate more use of that particular coping strategy.
Time Frame: up to 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Mediation Analysis (Symptom Burden and Coping) as Mediators of Improvement in Patient-reported QOL
Description: mediation analysis (mediation analyses are common in these types of studies, there is no novel new outcome measure here, but rather examining mediation)
Time Frame: 2 week
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Moderation Analysis to Examine Whether Patient or Transplant Related Characteristics Are Moderators of the Effect of the Intervention on Patient-reported QOL
Description: moderation analysis (moderation analyses are common in these types of studies. there is no new novel outcome measure here, bur rather examining moderation)
Time Frame: 2 week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 months after enrollment
Description: Given that this is a supportive care study, the protocol a priori specified that only averse events that are related to the study intervention or treatment would be reported. This is standard for supportive care trial in high-risk population where outcomes such as hospitalization/death are expected, but are not related to the study. That is how adverse events were defined and reported in this trial.
Groups:
- Inpatient Palliative Care Intervention Patient: * Patients will complete baseline self-report assessments at the time of obtaining informed consent
  * Patients will receive the palliative care intervention, which entails having twice weekly visits during the transplant hospitalization.
- Transplant Care Alone Patient: * Patients will complete baseline self-report assessments at the time of obtaining informed consent.
  * Standard Transplant Care
  Standard Transplant Care: Standard care per hospital guidelines
- Inpatient Palliative Care Intervention Caregiver: - Patients who enroll in the study may identify a caregiver to participate in the trial. The caregiver will follow the randomization of the patient. Caregivers of patients randomized to the palliative care intervention may meet with the palliative care clinicians during the patient's hospitalization for stem cell transplantation
- Transplant Care Alone Caregivers: -patients who enroll in the study may identify a caregiver to participate in the trial. The caregiver will follow the randomization of the patient. Caregivers of patients randomized to transplant care alone will receive usual transplant care per hospital guidelines.
Arm/Group | Inpatient Palliative Care Intervention Patient | Transplant Care Alone Patient | Inpatient Palliative Care Intervention Caregiver | Transplant Care Alone Caregivers
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/180 | 0/101 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180 | 0/101 | 0/85
Other Adverse Events (participants affected / at risk) | 0/180 | 0/180 | 0/101 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT03641378/Prot_SAP_000.pdf